CLINICAL TRIAL: NCT05984940
Title: Clinical Outcome of Root Canal Treatment With Ortho MTA (BioMTA®) Cement and AH Plus® Bioceramic Sealer (Dentsply). A Randomized Controlled Trial.
Brief Title: Treatment Outcome of Ortho MTA (BioMTA®) Cement vs AH Plus® Bioceramic Sealer (Dentsply).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/00168
Record Dates: First submitted 2023-07-12; First posted 2023-08-09 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2023-09

CONDITIONS: Endodontic Disease
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP and AH Plus sealer (Active Comparator): Root canal obturation using gutta percha and AH Plus® bioceramic sealer.
  Interventions: Device: GP and AH Plus sealer
- Ortho MTA (Experimental): Root canal obturation using Ortho MTA cement.
  Interventions: Device: Ortho MTA cement

INTERVENTIONS:
Device: Ortho MTA cement — Ortho MTA has a fine granularity for only 2 microns. It penetrates into dental tubules and fuses itself to the surface where it is applied. In addition, it prevents micro-leakage by forming an interfacing layer of hydroxyapatite (Hap) between the OrthoMTA and the canal wall.
  Arms: Ortho MTA
Device: GP and AH Plus sealer — AH Plus Sealer is a calcium silicate-based root canal sealer. Tricalcium Silicate interacts with body fluids to release calcium and hydroxide ions that promote hydroxyapatite (HA) formation.
  Arms: GP and AH Plus sealer

SUMMARY:
The use of bioceramics materials as root canal fillings in endodontics is gaining traction due to their excellent biocompatibility, antibacterial and sealing abilities. They are dispensed in the form of sealers and cements to be used with gutta-percha or mixed with liquids to form a paste. Recently, Ortho MTA (BioMTA®) cement is clinically available as a root filling material, without the need for gutta-percha. The purpose of this randomized controlled clinical trial is to compare clinical outcome between the novel Ortho MTA (BioMTA®) and the conventional gutta-percha with bioceramic sealer, when used as obturating materials in root canal treatment. This research aims to compare the healing outcome of infected teeth treated by root canal treatment and root-filled using MTA cement (Ortho MTA, BioMTA® Seoul Korea) or bioceramic sealer (AH Plus® Bioceramic Sealer (Dentsply).

The sealer can be used alone or in combination with gutta-percha obturating cones, injected gutta-percha material or core-carriers master cones. In vitro studies have demonstrated the capability of MTA to generate hydroxyapatite precipitates that penetrate into dentinal tubules.

DETAILED DESCRIPTION:
The use of bioceramics materials as root canal fillings in endodontics is gaining traction due to their excellent biocompatibility, antibacterial and sealing abilities. They are dispensed in the form of sealers and cements to be used with gutta-percha or mixed with liquids to form a paste.

In the sealer form, comparisons have been made between bioceramic and conventional resin-based sealers to study post-operative pain, cytocompatibility and bioactivity potential and treatment outcomes. In the cement form (MTA and Biodentine), they are largely used in apexification, regeneration endodontics, perforation repairs and apical surgeries. Recently, Ortho MTA (BioMTA®) cement is clinically available as a root filling material, without the need for gutta-percha. There are currently no systematic evaluations of this material therefore the purpose of this randomized controlled clinical trial is to compare clinical outcome between the novel Ortho MTA (BioMTA®) and the conventional gutta-percha with bioceramic sealer, when used as obturating materials in root canal treatment.

Mineralized Trioxide Aggregate (MTA) is a powder of fine trioxides (tricalcium oxides, silicon oxide, bismuth oxide) and hydrophilic particles (tricalcium silicate and tricalcium aluminate). It has good biocompatibility, antibacterial, dimensionally stable, provides hermetic seal against leakage and capable of stimulating healing and osteogenesis (bioactive). It is usually mixed with distilled water or saline to form colloidal gel with pH 12.5 and solidifies in 3-4 hours. The release of calcium hydroxide during setting are responsible for the high alkalinity, antibacterial and bioactivity.

Ortho MTA (BioMTA®) is an orthograde root canal filling material that was synthesized by mineral trioxide aggregate's active ingredient through Bio-ceramic manufacturing process. It was formulated to meet the ideal requirements of root canal filling material necessary for a clinically effective root canal treatment on cases of file separation, cracked tooth, severely infected canal, and treatment of acute apical abscess. It is packaged as powder in a vial and mixed with distilled water where setting begins and continues in vivo.

AH Plus® Bioceramic Sealer is a root canal sealer conforming to ISO 6876, in a pre-loaded syringe that does not require any pre-mixing and is set by absorbing moisture from the root canal environment. The sealer can be used either alone or in combination with gutta-percha obturating cones, injected gutta-percha material or core-carriers master cones.

Root canal treatment often uses gutta-percha and sealers to provide 3-dimensional hermetic seal of a cleaned and disinfected canal. To date, studies exploring root canal treatment with bioceramic and resin-based sealers have showed comparable results. At the same time, MTA has been widely used over the past 30 years in a variety of endodontic treatment targeted at restoring compromised teeth, including as apical barriers/seals for immature tooth with open apices, in root end surgeries root perforation repairs, preservation of the carious vital pulp and revitalization of infected immature teeth. Especially among teeth weakened by infection, the concept of a "monoblock" of root canal filling that is bonded to dentine to strengthen the tooth, is attractive. While clinical research into the monoblock root filling created by conventional gutta-percha and sealer has failed to show significant advantage, in vitro studies have demonstrated the capability of MTA to generate hydroxyapatite precipitates that penetrate into dentinal tubules, taking the technology one step closer to the monoblock concept. Hence, the purpose of this research is to compare the healing outcome of infected teeth treated by root canal treatment and root-filled using MTA cement (Ortho MTA, BioMTA® Seoul Korea) or bioceramic sealer (AH Plus® Bioceramic Sealer (Dentsply).

ELIGIBILITY:
Inclusion Criteria:

* A preoperative periapical radiograph will be required for diagnosis.
* Subjects at least 21 years old to 95 years old.
* Medically healthy
* In a patient with multiple teeth requiring root canal treatment, only 1 tooth from each side will be included and selected at random.
* Tooth requiring root canal treatment presenting with periapical radiolucency.

Exclusion Criteria:

* Patients below 21 years old.
* Pregnant women.
* Patients with autoimmune disease and uncontrolled diabetes.
* Teeth with periodontal probing depth 5mm or more.
* Incomplete root formation that is detected radiographically.
* Cracked teeth.
* Teeth are deemed to have poor restorative prognosis.
* Teeth with adjacent teeth on the same side that require root canal treatment.

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Objectives (Change in baseline periapical lesion size at 6 month and 12 month) | 6, 12 months
  Change in baseline periapical lesion size at 6 month and 12 month

SECONDARY OUTCOMES:
Secondary Objectives (Change in baseline post-operative pain at Day 1, Day 3 and Day 7 post treatment) | 1, 3, 7 days
  Change in baseline post-operative pain at Day 1, Day 3 and Day 7 post treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No